CLINICAL TRIAL: NCT05584982
Title: Open-label, Single-arm, Investigator-Initiated Clinical Study to Investigate the Performance of the AtbFinder® Diagnostic Test System for Selection of Antibiotic Therapy in Persons With Cystic Fibrosis
Brief Title: Clinical Performance of the AtbFinder® Test System for Selection of Antibiotic Therapy in Persons With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TGV-Dx (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Atbfinder-CF1
Record Dates: First submitted 2022-10-12; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Cystic Fibrosis; Lung Infection Bacterial
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AtbFinder-1 (Experimental): persons with cystic fibrosis to whom AtbFinder was used to formulate an individualized antibiotic regimen
  Interventions: Device: AtbFinder

INTERVENTIONS:
Device: AtbFinder — In the present study, we provided a prospective evaluation of the effectiveness of antibiotics selected with AtbFinder compared to a retrospective analysis of antibiotic efficacy selected with conventional culture-based antibiotic susceptibility tets in patients with cystic fibrosis

SUMMARY:
This prospective case-control study was planned to evaluate the efficacy of antibiotic therapy selected with the AtbFinder® in persons with cystic fibrosis.

DETAILED DESCRIPTION:
This pilot study entitled "Clinical Performance of the AtbFinder® diagnostic test system for selection of antibiotic therapy in persons with cystic fibrosis " was designed to demonstrate the clinical performance of antibiotics selected with the AtbFinder® for the treatment of lung infections in persons with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis based on sweat chloride levels = or > 60, or genetic testing showing 2 pathogenic mutations.
* Ability to provide a clinical sample (expectorated sputum, throat culture or bronchoalveolar lavage) prior to the start of the antibiotic treatment.
* Prior treatment of a pulmonary exacerbation with systemic antibiotics in the preceding year.

Exclusion Criteria:

* Inability to meet any of the above inclusion criteria.
* Systemic therapy with an antibiotic or corticosteroids in the 3 weeks preceding enrollment in the study, except those on chronic inhaled antibiotics.
* Primary or secondary (drug- or condition-induced) immune compromise.
* Creatinine > 2 x upper limit of normal for age.
* Previous participation in this study in the prior 28 days.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-01; Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Time to an exacerbation (in months) | Time Frame: up to 24 months

SECONDARY OUTCOMES:
Evaluate changes in forced expiratory volume from baseline to end of study | Time Frame: up to 24 months
Changes in Pseudomonas aeruginosa load (the number of colony forming units per 1 ml of sputum) from baseline to end of treatment | Time Frame: up to 24 months
Changes in bacterial load of isolated organisms (the number of colony forming units per 1 ml of sputum) from baseline to end of treatment | Time Frame: up to 24 months
Changes in blood white blood cell count (10*9 mg/L) | Time Frame: up to 24 months
Changes in blood C-reactive protein (in mg/L) | Time Frame: up to 24 months
Changes in weight (in kilograms) | Time Frame: up to 24 months
Changes in body mass index calculated as weight (in kilograms) divided by height squared (m2). | Time Frame: up to 24 months

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 2022-2023